CLINICAL TRIAL: NCT04679259
Title: Evaluation of Blood Biomarkers as an Indicator of Delayed Neurocognitive Recovery After Cardiac Surgery
Brief Title: Evaluation of Blood Biomarkers as an Indicator of Delayed Neurocognitive Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, Associate professor, SMG-SNU Boramae Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 30-2020
Record Dates: First submitted 2020-12-11; First posted 2020-12-22 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2020-12

CONDITIONS: Postoperative Cognitive Dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac surgical patients (Experimental)
  Interventions: Diagnostic Test: Blood sampling for assessment of the level of D-Amino Acid Oxidase, D-serine and Serine in blood; Diagnostic Test: Neurocognitive test; Diagnostic Test: Assessment of delirium

INTERVENTIONS:
Diagnostic Test: Blood sampling for assessment of the level of D-Amino Acid Oxidase, D-serine and Serine in blood — Blood sampling is done before surgery and at 1, 2, and 7 day after surgery. The level of D-Amino Acid Oxidase, D-serine and Serine in blood are assessed.
Diagnostic Test: Neurocognitive test — Neurocognitive test is performed before surgery and at 7 day after surgery
Diagnostic Test: Assessment of delirium — Postoperative delirium is assessed daily during 7 days after surgery.

SUMMARY:
Delayed neurocognitive recovery is defined as a cognitive decline arising after surgery. In the present study, the authors evaluate the level of D-Amino Acid Oxidase, D-serine and Serine racemase in blood as an indicator of delayed neurocognitive recovery after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective cardiac surgery

Exclusion Criteria:

* MMSE <24
* History of psychological or neurological diseases
* Illiteracy
* Preoperative delirium
* Vision and hearing impairment

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Change of concentration of D-Amino Acid Oxidase in blood at 1, 2, and 7 day after surgery | Before surgery and at 1, 2, and 7 day after surgery
  Blood level of D-Amino Acid Oxidase is assessed.

SECONDARY OUTCOMES:
Concentration of D-serine in blood | Before surgery and at 1, 2, and 7 day after surgery
  Blood level of D-serine is assessed.
Concentration of Serine racemase in blood | Before surgery and at 1, 2, and 7 day after surgery
  Blood level of Serine is assessed.
Occurrence of delayed neurocognitive recovery | Before surgery and at 7 day after surgery
  Neurocognitive assessment

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Select State/Province, South Korea

IPD SHARING:
Plan to Share IPD: Undecided